CLINICAL TRIAL: NCT04391010
Title: Effectiveness of Respirators Fit Factor in Healthcare Providers With and Without Beard: A Randomized Clinical Trial
Brief Title: Effectiveness of Respirators Fit Factor in Healthcare Providers With and Without Beard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UCM Respirators Fit Factor
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Community Health Workers; Filtration; Masks
MeSH Terms: interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health care providers with beard (Other)
  Interventions: Other: Surgical masks; Other: Filtering respirators
- Health care providers without beard (Other)
  Interventions: Other: Surgical masks; Other: Filtering respirators

INTERVENTIONS:
Other: Surgical masks — Surgical masks will be applied in health care providers
Other: Filtering respirators — Filtering respirators will be applied in health care providers

SUMMARY:
The study aim will be to determine the fit factor of surgical masks and filtering respirators in healthcare providers with and without beard. A randomized clinical trial will be carried out recruiting a sample of 52 healthcare providers with and without beard. Fit factor will be measured with both surgical masks and filtering respirators and compared between healthcare providers with and without beard.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers

Exclusion Criteria:

* Pulmonary diseases
* Pregnant women
* Not sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Fit factor | Change from baseline fit factor immediately after intervention
  Particles count into masks compared to particles count outside of the masks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No